CLINICAL TRIAL: NCT00705198
Title: Temodal Capsule All-Case-Registered Surveillance (Designated Drug Use Investigation) - Evaluation of The Safety and Efficacy of Temodal in Patients With Newly Diagnosed Malignant Glioma (Concomitant With Radiotherapy and Then as Monotherapy) and Relapsed Malignant Glioma (as Monotherapy)
Brief Title: Temozolomide All-Case-Registered Surveillance (Designated Drug Use Investigation)(Study P05062)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05062
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Glioma; Astrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Newly diagnosed patients: Patients treated with temozolomide for newly diagnosed malignant glioma
  Interventions: Drug: Temozolomide (for newly diagnosed malignant glioma); Radiation: Radiotherapy (for patients with newly diagnosed malignant glioma)
- Relapsed patients: Patients treated with temozolomide for relapsed malignant glioma
  Interventions: Drug: Temozolomide (for relapsed malignant glioma)
- Newly diagnosed anaplastic astrocytoma patients: Patients treated with temozolomide for newly diagnosed anaplastic astrocytoma
  Interventions: Drug: Temozolomide (for newly diagnosed malignant glioma); Radiation: Radiotherapy (for patients with newly diagnosed malignant glioma)

INTERVENTIONS:
Drug: Temozolomide (for newly diagnosed malignant glioma) — Temozolomide treatment for newly diagnosed malignant glioma. The usual dose for adults in combination with radiotherapy is 75 mg/m2 orally once daily for 42 consecutive days. After a 4 week rest period, monotherapy at 150 mg/m2 orally once daily for 5 consecutive days per 28 day treatment cycle is administered. The dose may be increased to 200 mg/m2 for the next 28 day treatment cycle.
  Temozolomide is administered as 20 mg and 100 mg capsules.
  Other Names: Temodal; Temodar; SCH 052365
  Groups: Newly diagnosed anaplastic astrocytoma patients; Newly diagnosed patients
Drug: Temozolomide (for relapsed malignant glioma) — Temozolomide treatment for relapsed malignant glioma. The usual dose for adults is 150 mg/m2 orally once daily for 5 consecutive days per 28 day treatment cycle. The dose may be increased to 200 mg/m2 for the next 28 day treatment cycle.
  Temozolomide is administered as 20 mg and 100 mg capsules.
  Other Names: Temodal; Temodar; SCH 052365
  Groups: Relapsed patients
Radiation: Radiotherapy (for patients with newly diagnosed malignant glioma) — Although the study protocol does not clearly define how long this intervention is applied, radiotherapy is generally administered 5 days/week for 6 weeks to patients with newly diagnosed malignant glioma.
  Other Names: Radiation therapy
  Groups: Newly diagnosed anaplastic astrocytoma patients; Newly diagnosed patients

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of temozolomide in patients with newly diagnosed malignant glioma (concomitant with radiotherapy and then as monotherapy) and relapsed malignant glioma (as monotherapy) when used in the daily medical practices.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

DETAILED DESCRIPTION:
Patients are invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with temozolomide for newly diagnosed malignant glioma (concomitant with radiotherapy and then as monotherapy) and relapsed malignant glioma (as monotherapy).

Exclusion Criteria:

* Patients with a history of hypersensitivity to temozolomide or dacarbazine.
* Pregnant women and women who may be pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with temozolomide for newly diagnosed malignant glioma (concomitant with radiotherapy and then as monotherapy) and relapsed malignant glioma (as monotherapy). In addition, up to 450 patients with newly diagnosed anaplastic astrocytoma will be registered to investigate survival time.
Sampling Method: Non-Probability Sample
Enrollment: 1804 (Actual)
Dates: Start 2006-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety: observation of hematology, biochemistry, and adverse events (AEs); evaluation of details of occurrence of AEs and unexpected serious AEs, and evaluation of presence or absence of secondary malignancies and causal relationship with temozolomide. | AEs during treatment with temozolomide, serious AEs occurring within 30 days after completion of treatment with temozolomide. Secondary malignancies will be monitored from the start of treatment with temozolomide to final outcome.
Efficacy in patients registered during Period 1, evaluated as Remarkably Effective, Moderately Effective, Stable Disease, Progression, or Not Evaluable, considering tumor responses, progression free survival, overall survival, among other factors. | One year after start of temozolomide treatment.
Efficacy in all newly diagnosed anaplastic astrocytoma patients:, evaluated as 5 year survival rate and overall survival. | From the start of treatment with temozolomide to final outcome.